CLINICAL TRIAL: NCT06833658
Title: Effects of Aromatherapy with Essential Oils on Anxiety and Depression in Perioperative Patients with Pancreatic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023yan540-002
Record Dates: First submitted 2024-12-12; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Carcinoma
Keywords: Aromatherapy with essential oil intervention; pancreatic carcinoma; Anxiety; Depression
MeSH Terms: conditions — Pancreatic Neoplasms; Anxiety Disorders; Depression | interventions — Control Groups; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients should complete the self-rating Anxiety Scale (SAS) and Self-rating Depression Scale (SDS) within 24 hours on the day of admission. If the preoperative SAS score is ≥50 or (and)SDS score is ≥53, they can participate in this project, and then you need to sign the informed consent. According to the inclusion and exclusion criteria and admission to ward 1 and Ward 2, they were divided into test group and control group. The general information questionnaire was completed within 24 hours on the day of admission. Patients in ward 2 were given routine treatment, and patients in ward 1 selected several essential oils, diluted with tap water and scented with an aromatherapy machine, 1h each time, once in the afternoon. The intervention lasted a total of 15 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aromatherapy with essential oil intervention (Experimental): The 15-day intervention commenced one day prior to surgery and concluded on the 13th post-operative day. Psychological support was delivered through bedside face-to-face interviews with patients. Aromatherapy, customized to meet the psychological needs of pancreatic cancer patients, was employed as part of the intervention. A senior aromatherapist developed the protocol, selecting pleasant essential oils diluted at a ratio of 1-2 drops in 70ml of water. The aromatherapy was administered twice daily for one hour each session using an aromatherapy diffuser.During aromatherapy, nurses should inspect patients every 30 minutes to ensure comfort, and take immediate action if discomfort is reported. Prior to surgery, patients complete anxiety and depression self-assessment scales on the 14th and 42nd days post-operation. If discharged early, a telephone follow-up with a nurse on the 42nd day is conducted to complete the assessment.
  Interventions: Other: Experimental: Aromatherapy with essential oil intervention
- control group (Placebo Comparator): The control group offers high - quality and personalized nursing care to patients in line with the "High - quality Nursing Service" principles. The care details are as follows:
  1. Pre - operation: Present pancreatic cancer knowledge, such as causes, common symptoms, treatment methods, and the need for surgery. Answer patients' queries promptly to reduce their fear of the disease and surgery.
  2. Post - operation: Report the surgical outcome, explain common post - op complications and solutions to relieve negative emotions.
  3. Post - operation: Intensify post - op education on drainage tube care, activity guidelines, disease knowledge, and diet advice. Strengthen mental health education, encourage family members to show more concern for patients, and enhance family support.
  4. Pre - discharge: Provide discharge instructions to patients and their families. Guide patients who need tube removal and suture removal after discharge to make online appointments for outpatient follow - up.
  Interventions: Other: Control Group 0.9% Isotonic Saline

INTERVENTIONS:
Other: Experimental: Aromatherapy with essential oil intervention — Aromatherapy, customized to meet the psychological needs of pancreatic cancer patients, was employed as part of the intervention. A senior aromatherapist developed the protocol, selecting pleasant essential oils diluted at a ratio of 1-2 drops in 70ml of water. The aromatherapy was administered twice daily for one hour each session using an aromatherapy diffuser.During aromatherapy, nurses should inspect patients every 30 minutes to ensure comfort, and take immediate action if discomfort is reported.
  Other Names: Essential oil aromatherapy
  Arms: Aromatherapy with essential oil intervention
Other: Control Group 0.9% Isotonic Saline — 1. Pre - operation: Present pancreatic cancer knowledge, such as causes, common symptoms, treatment methods, and the need for surgery. Answer patients' queries promptly to reduce their fear of the disease and surgery. 2. Post - operation: Report the surgical outcome, explain common post - op complications and solutions to relieve negative emotions. 3. Post - operation: Intensify post - op education on drainage tube care, activity guidelines, disease knowledge, and diet advice. Strengthen mental health education, encourage family members to show more concern for patients, and enhance family support. 4. Pre - discharge: Provide discharge instructions to patients and their families. Guide patients who need tube removal and suture removal after discharge to make online appointments for outpatient follow - up.
  Arms: control group

SUMMARY:
The objective of this study is to investigate whether aromatherapy essential oils are effective in alleviating anxiety and depression in participants undergoing perioperative pancreatic cancer treatment. Researchers compared aromatherapy essential oils with a placebo (a substance that appears similar but contains no essential oils) to determine their efficacy in reducing anxiety and depression in these participants. Participants were required to undergo aromatherapy for 2 hours daily over a period of 15 days. Assessments of anxiety and depression were conducted one day before surgery, 14 days after surgery, and 42 days after surgery, with their scores recorded accordingly.

DETAILED DESCRIPTION:
Female participants in this study must not be pregnant or breastfeeding during the project period. Although the essential oils used in aromatherapy have minimal effects on infants, there remains a slight risk of developmental issues. Therefore, participants are required to use contraception. If pregnancy occurs or is suspected during the study period, the participant must immediately notify the researcher to terminate their participation and receive further guidance. Male participants are also required to use contraception.Participation in this study is entirely voluntary and free of charge. You may choose not to participate or withdraw at any time, and this will not have any adverse effects on your medical care. If you decide to withdraw, please promptly inform your study physician to obtain relevant health advice. We will also promptly inform you of any significant information that may affect your decision to participate.Regulatory authorities may decide to terminate the study during the research period. If the study is concluded prematurely, we will notify you immediately, and your study physician will provide recommendations for subsequent treatment based on your health condition. If you choose to withdraw from the study midway, we will offer a final follow-up, but you have the option not to participate. After withdrawing from the study, if there is new information concerning your health and rights, we may contact you. Following your withdrawal, your information will be kept strictly confidential until its destruction and will not be further used or disclosed. However, in certain exceptional circumstances, even after your withdrawal or the conclusion of the study, researchers may still use or disclose your information.Unless it affects the scientific integrity of the research or the evaluation of data security, your information will not be disclosed; only information necessary for research, teaching, and other related activities will be provided, excluding personal identification details such as names and ID numbers. If required by government regulatory authorities, all research information, including your participation details, will be provided.If participation in this study results in any health impairment, please contact the researchers (Liu Xiaoyi, 83572652) immediately. We will promptly provide necessary medical treatment and offer compensation in accordance with national legal regulations.Your personal information and participation in this study will be strictly confidential and will not be disclosed to anyone outside the research team without authorization. All researchers are obligated to protect your privacy. Your data will be stored in a locked file cabinet and will only be accessible to authorized researchers. To ensure compliance with research regulations, government or ethics committee members may need to review your information. When the research results are published, your personal data will not be disclosed.If you have any questions regarding the rights and interests of the participants, you may contact the Biomedical Research Ethics Committee of Peking University First Hospital at the following telephone number: 010-66119025.

Informed Consent Signature Page Subject's Informed Consent Statement The researcher has explained to me the background, purpose, procedures, risks, and benefits of the study titled "The Effect of Aromatherapy Essential Oils on Anxiety and Depression in Perioperative Pancreatic Cancer Participants." I have had sufficient time and opportunity to ask questions, and I am satisfied with the answers provided by the researcher. I know whom to contact if I have further questions or need additional information. I have read this informed consent form and decided to participate in this study. I understand that I may withdraw from this study at any time during the research period without providing any reason. I have been informed that I will receive a copy of this informed consent form, which includes both my signature and the researcher's signature.

Subject's Signature: ___________________________ Date: _______________

Researcher's Declaration I have explained to the subject the background, purpose, procedures, risks, and benefits of the study titled "The Effect of Aromatherapy Essential Oils on Anxiety and Depression in Perioperative Pancreatic Cancer Participants." I have provided sufficient time for the subject to read the informed consent form, discuss it with others, and have answered all questions regarding the study. I have informed the subject of the contact information for any research-related inquiries. I have also informed the subject that they may withdraw from the study at any time without providing any reason.

Researcher's Signature: ___________________________ Date: _______________

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria in Chinese Anti-Cancer Association Guidelines for pancreatic cancer
* Age ≥18 years
* Contraception required, non-lactation period
* Consistent with surgical indications
* Surgical procedures: pancreaticoduodenectomy, extended pancreaticoduodenectomy, costocaudectomy, total pancreatectomy, subtotal pancreatectomy, pyloric-sparing pancreaticoduodenectomy
* Elective surgery without preoperative radiotherapy or chemotherapy
* Normal communication
* Preoperative SAS score ≥50 or SDS score ≥53
* Informed consent from subject or guardian

Exclusion Criteria:

* History of mental illness or cognitive impairment
* Severe liver/kidney disease, cardiopulmonary dysfunction, tumor recurrence/metastasis
* Allergy or intolerance to aromatic reagents, olfactory disorders, acute respiratory disease, serious complications (unstable vital signs, blood clotting disorders, irreversible metabolic diseases)
* Poor compliance with study protocol or participation in similar studies
* Termination due to disease treatment or condition changes
* Withdrawal for personal reasons
* Deemed unsuitable by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Self-rating Anxiety Scale (SAS) | Within 24 hours on the day of admission, after intervention (14 days after surgery) and 28 days after intervention (42 days after surgery).
  Zung[20] self-rating Anxiety Scale was adopted, which was compiled in 1971, with a total of 20 items, and scored according to the four levels of "no or occasionally (1 point)","sometimes (2 points)", "often (3 points)" and"always (4 points) ", in which items 5, 9, 13, 17 and 19 were scored in reverse. Add the scores of all items, multiply by the coefficient 1.25, and take their integer parts and remember them to the standard score. After the Chinese revision of the scale in China, the norm results are judged as follows: SAS standard score <50 is no anxiety, 50 ~ 59 is mild anxiety, 60 ~69 is moderate anxiety, ≥70 is severe anxiety, the higher the score, the more serious the anxiety. Cronbach's a coefficient of the scale was 0.799, indicating good reliability and validity.
Self-rating Depression Scale (SDS) | Within 24 hours on the day of admission, after intervention (14 days after surgery) and 28 days after intervention (42 days after surgery).
  The Zung[21] Self-rating Depression Scale, which was developed in 1965, was used to assess the subjective feelings of individuals with depressive symptoms. There are 20 items that are scored on a 4-point scale based on the frequency of symptoms, where "1" means no or occasionally, "2" means sometimes, "3" means often, and "4" means always. Items 2, 5, 6, 11, 12, 14, 16, 17, 18, and20 are negative scoring questions, which are calculated as 4 to 1 points. Add the scores of all items, multiply by the coefficient1.25, and take their integer parts and remember them to the standard score. A standard score of <53 indicates no depression, a score of 53-62 indicates mild depression, a score of 63-72 indicates moderate depression, a score of ≥73 indicates severe depression, and the higher the score, the more severe the depression. Cronbach's a coefficient of this scale was 0.78, indicating good reliability and validity.

IPD SHARING:
Plan to Share IPD: No